CLINICAL TRIAL: NCT00444106
Title: An Open-label, Randomized, Single-center, Parallel Group Study of the Effects of Artemether-lumefantrine (Coartem®) Atovaquone-proguanil (Malarone®) and Artesunate-mefloquine on Auditory Function Following the Treatment of Acute Uncomplicated Plasmodium Falciparum Malaria in Patients 12 Years of Age or Older
Brief Title: Evaluation of Potential Effect of Artemether - Lumefantrine and Malaria Drugs on Auditory Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCOA566A2417
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Results first posted 2011-03-16 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Malaria; Falciparum
Keywords: Malaria; hearing; co-artemether; auditory; Plasmodium falciparum; marsh fever; Plasmodium infections; remittent fever; paludism; artemether; artemisinins; benflumetol; lumefantrine
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Mefloquine; atovaquone, proguanil drug combination; Artemether, Lumefantrine Drug Combination

ARMS (3):
- Artemether-lumefantrine (Coartem) (Experimental): Artemether-lumefantrine (Coartem) tablets containing 20 mg artemether and 120 mg lumefantrine twice a day for 3 days, dosage dependent on body weight.
  Interventions: Drug: Artemether-lumefantrine
- Atovaquone-proguanil (Malarone) (Active Comparator): Atovaquone-proguanil (Malarone) tablets containing 250 mg atovaquone and 100 mg proguanil hydrochloride once daily for 3 days, dosage dependent on body weight.
  Interventions: Drug: Atovaquone-proguanil
- Artesunate-mefloquine (Active Comparator): Artesunate-mefloquine tablets containing 50 mg artesunate (Plasmotrim) and 250 mg mefloquine (Mephaquin). Artesunate 4 mg/kg/day (for 3 days) and mefloquine 25 mg/kg/day (days 2 and 3) total dose was given once daily dependent upon body weight.
  Interventions: Drug: Artesunate-mefloquine

INTERVENTIONS:
Drug: Artesunate-mefloquine
  Other Names: Plasmotrim; Mephaquin
  Arms: Artesunate-mefloquine
Drug: Atovaquone-proguanil
  Other Names: Malarone
  Arms: Atovaquone-proguanil (Malarone)
Drug: Artemether-lumefantrine
  Other Names: Coartem
  Arms: Artemether-lumefantrine (Coartem)

SUMMARY:
To evaluate the potential effects of artemether- lumefantrine on the auditory function

ELIGIBILITY:
Inclusion Criteria

* 12 years of age or older
* Accepts Healthy Volunteers
* P. falciparum parasitemia between 1,000 and 100,000 parasites/μl
* History of fever or presence of fever (temperature ≥ 37.5°C)

Exclusion Criteria

* Signs/symptoms of severe/complicated malaria
* Ingestion of various antimalarial drugs, or antibiotics in the previous 2 weeks to 2 months
* History of any drug-related hearing impairment
* Abnormal hearing function at study entry
* Exposure to sustained loud noises, by self-report, within the past 24 hours
* Present ear problems
* Pregnant or lactating (urine test for β-HCG) to be performed on any woman of child bearing age)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2007-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis Investigational Site, Tumaco, Colombia

RESULTS

PARTICIPANT FLOW:
Groups:
- Artemether-lumefantrine (Coartem): Artemether-lumefantrine (Coartem) tablets containing 20 mg artemether and 120 mg lumefantrine twice a day for 3 days dosage dependent on body weight.
- Atovaquone-proguanil (Malarone): Atovaquone-proguanil (Malarone) tablets containing 250 mg atovaquone and 100 mg proguanil hydrochloride once daily for 3 days dosage dependent on body weight.
- Artesunate-mefloquine: Artesunate (Plasmotrim) 50 mg tablet; based on body weight for a dosage of 4 mg/kg/day for 3 days- mefloquine (Mephaquin) 250 mg tablets; based on body weight for a total dosage of 25 mg/kg once daily on days 2 and 3.
Period: Overall Study
Arm/Group | Artemether-lumefantrine (Coartem) | Atovaquone-proguanil (Malarone) | Artesunate-mefloquine
Started | 159 | 53 | 53
Completed Treatment Period | 159 | 53 | 53
Completed | 157 | 52 | 52
Not Completed | 2 | 1 | 1
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Abnormal Test Procedure Results | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Artemether-lumefantrine (Coartem) | Atovaquone-proguanil (Malarone) | Artesunate-mefloquine | Total
Number analyzed (Participants) | 159 | 53 | 53 | 265
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 51 | 21 | 18 | 90
  Between 18 and 65 years | 108 | 32 | 35 | 175
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.6 (11.6) | 25.1 (11.16) | 25.2 (11.26) | 25.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 19 | 22 | 104
  Male | 96 | 34 | 31 | 161
Body Weight [Mean (Standard Deviation); unit: kg] | 62.8 (14.39) | 60.3 (14.54) | 65.2 (15.37) | 62.8 (14.64)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Auditory Abnormalities at Day 7 Assessed by Auditory Brainstem Response (ABR) Wave III Latency Changes on Day 7(a Type of Hearing Test)
Description: To demonstrate the safety of artemether-lumefantrine after 3 days of treatment in patients with acute, uncomplicated falciparum malaria by testing the null hypothesis that the rate of auditory abnormalities is ≥ 15% in the population treated with artemether-lumefantrine as assessed by ABR at Day 7 following initiation of treatment compared with their baseline values. An "auditory nerve abnormality" is here defined as a greater than 0.30 ms change in Wave III latency from baseline to Day 7. Exact Pearson-Clopper two-sided 95% confidence limits were constructed for all three treatment groups.
Time Frame: 7 days
Population: Safety per protocol set defined as all the randomized patients who took at least 80% of the entire recommended dose and had a valid baseline and Day 7 ABR Wave III latency evaluation and did not use any meds having an ototoxic effect.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Artemether-lumefantrine (Coartem)
Number analyzed (Participants) | 151
Percentage of Participants | 2.6 [0.7 to 6.6]
Statistical Analysis 1: Comparison: Artemether-lumefantrine (Coartem); One-sided null hypothesis that the incidence rate of ABR Wave III latency changes is greater than or equal to 15%. Increase in ABR Wave III latency between baseline and Day 7 of greater than 0.3 ms; Test type: Superiority or Other; p < .0001, One-sided exact test for a single propn; One-sided exact test for a single proportion

2. Secondary Outcome: Auditory Changes Following 3 Days of Treatment at Days 3, 7, 28, and 42 Days as Assessed by Pure Tone Thresholds Assessments (a Type of Hearing Test)
Description: Audiometric measurements such as pure-tone threshold (air conduction tested at 250 to 8000 HZ) day 3, 7, 28 and 42 following initiation of treatment, including changes from baseline. Pure-tone average (PTA) calculated for each ear by averaging the pure-tone threshold values at 500, 1000, 2000 and 3000 HZ.
Time Frame: Baseline (Day 1), 3, 7, 28 and Day 42
Population: Safety per protocol patients who had a valid ABR at baseline and on the specified day were included.
Measure: Mean (95% Confidence Interval); unit: dB
Groups:
- Artemether-lumefantrine: Artemether-lumefantrine (Coartem) tablets containing 20 mg artemether and 120 mg lumefantrine twice a day for 3 days dosage dependent on body weight.
- Atovaquone-proguanil (Malarone): Atovaquone-proguanil (Malarone) 250mg tablets once daily for 3 days dosage dependent on body weight.
- Artesunate-mefloquine: Artesunate (Plasmotrim) 50 mg tablet; based on body weight for a dosage of 4 mg/kg/day for 3 days- mefloquine (Mephaquin)250 mg tablets; based on body weight for a total dosage of 25 mg/kg once daily on days 2 and 3.
Arm/Group | Artemether-lumefantrine | Atovaquone-proguanil (Malarone) | Artesunate-mefloquine
Number analyzed (Participants) | 148 | 51 | 47
dB
  Baseline Right Ear | 12.2 [11.4 to 13.0] | 12.0 [10.5 to 13.6] | 12.7 [11.2 to 14.2]
  Change from baseline to Day 3 Right Ear | -2.5 [-3.1 to -1.9] | -2.4 [-3.6 to -1.2] | -1.9 [-3.0 to -0.7]
  Change from baseline to Day 7 Right Ear | -2.2 [-2.9 to -1.5] | -2.6 [-4.0 to -1.1] | -2.6 [-3.9 to -1.3]
  Change from baseline to Day 28 Right Ear | -2.7 [-3.5 to -1.9] | -2.6 [-4.2 to -1.0] | -3.6 [-4.8 to -2.3]
  Change from baseline to Day 42 Right Ear | -3.0 [-3.8 to -2.2] | -3.3 [-4.9 to -1.7] | -3.1 [-4.2 to -1.9]
  Baseline Left Ear | 11.4 [10.5 to 12.3] | 11.3 [9.9 to 12.7] | 12.5 [10.8 to 14.3]
  Change from baseline to Day 3 Left Ear | -1.2 [-1.8 to -0.5] | -1.5 [-2.6 to -0.3] | -1.2 [-2.2 to -0.1]
  Change from baseline to Day 7 Left Ear | -1.7 [-2.4 to -0.9] | -1.3 [-2.8 to 0.2] | -1.4 [-2.8 to -0.1]
  Change from baseline to Day 28 Left Ear | -2.0 [-2.8 to -1.1] | -1.8 [-3.0 to -0.5] | -2.5 [-4.3 to -0.7]
  Change from baseline to Day 42 Left Ear | -1.5 [-2.7 to -0.4] | -2.1 [-3.5 to -0.6] | -3.0 [-4.7 to -1.3]

3. Secondary Outcome: Relationship Between Changes in Auditory Function and Treatment Groups
Description: ABR Wave III latency (ms) changes from baseline to Day 7 in the three drug exposure groups.
Time Frame: From Baseline to Day 7
Measure: Mean (95% Confidence Interval); unit: ms
Arm/Group | Artemether-lumefantrine (Coartem) | Atovaquone-proguanil (Malarone) | Artesunate-mefloquine
Number analyzed (Participants) | 151 | 50 | 45
ms
  Baseline Right Ear | 3.86 [3.83 to 3.90] | 3.89 [3.84 to 3.94] | 3.86 [3.8 to 3.93]
  Change from baseline to Day 7 Right Ear | 0.01 [-0.01 to 0.03] | -0.01 [-0.04 to 0.02] | -0.04 [-0.08 to 0.01]
  Baseline Left Ear | 3.85 [3.82 to 3.88] | 3.88 [3.84 to 3.93] | 3.82 [3.77 to 3.88]
  Change from baseline to Day 7 Left Ear | 0.01 [-0.01 to 0.03] | -0.01 [-0.04 to 0.02] | -0.03 [-0.07 to 0.0]

4. Secondary Outcome: Efficacy of Polymerase Chain Reaction (PCR) Adjusted Malaria Cure Rates of the Three Treatment Regimens at Days 14, 28 and 42
Description: Percentage of patients with clearance of asexual parasitemia (observed by optical microscopy) within 7 days of initiation of trial treatment without recrudescence within 14, 28 and 42 days respectively after initiation of treatment. Patients with recurrent parasitemia and paired PCR results were classified as either a new infection (different paired genotypes) or a recrudescence (matching paired genotypes). Patients without paired PCR results or ambiguous results were classified as treatment failures.
Time Frame: Days 14, 28 and 42
Population: Full Analysis Set defined as all randomized patients with confirmed malaria at baseline, who had at least one dose of study drug and had at least one relevant post-baseline efficacy assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Artemether-lumefantrine (Coartem) | Atovaquone-proguanil (Malarone) | Artesunate-mefloquine
Number analyzed (Participants) | 151 | 53 | 53
Percentage of Participants
  Day 14 | 99.4 [96.5 to 100.0] | 100.0 [93.3 to 100.0] | 98.1 [89.9 to 100.0]
  Day 28 | 98.7 [95.5 to 99.8] | 98.1 [89.9 to 100.0] | 98.1 [89.9 to 100.0]
  Day 42 | 97.5 [93.7 to 99.3] | 98.1 [89.7 to 100.0] | 98.1 [89.9 to 100.00]

ADVERSE EVENTS:
Description: Safety Set- All patients who received at least one dose of study drug and had at least one post baseline safety assessment.
Groups:
- Artemether-lumefantrine: Artemether-lumefantrine
- Atovaquone-proguanil: Atovaquone-proguanil
- Artesunate-Mefloquine: Artesunate-Mefloquine
Arm/Group | Artemether-lumefantrine | Atovaquone-proguanil | Artesunate-Mefloquine
Serious Adverse Events (participants affected / at risk) | 0/159 | 0/53 | 1/53
Other Adverse Events (participants affected / at risk) | 23/159 | 17/53 | 30/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Artemether-lumefantrine (N=159) | Atovaquone-proguanil (N=53) | Artesunate-Mefloquine (N=53)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Artemether-lumefantrine (N=159) | Atovaquone-proguanil (N=53) | Artesunate-Mefloquine (N=53)
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 7
Vomiting (Gastrointestinal disorders) | 2 | 9 | 15
Pyrexia (General disorders) | 6 | 4 | 2
Dizziness (Nervous system disorders) | 9 | 5 | 14
Headache (Nervous system disorders) | 5 | 7 | 7
Insomnia (Psychiatric disorders) | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.